CLINICAL TRIAL: NCT02566005
Title: A Randomized Comparison of Transcervical Foley Bulb With Vaginal Misoprostol to Vaginal Misoprostol Alone for Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-0032
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy
Keywords: Misoprostol; Induction; Foley

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol group (Active Comparator): The women in the misoprostol only group will receive 25mcg of misoprostol per vagina every 4hours per the standard hospital protocol. Once the cervix becomes favorable or if the patient is in active labor, or if there is no progress for 24 hours, misoprostol administration will be discontinued. Further management of labor will depend on the labor team. (25mcg tablets are not available commercially; a 100mcg table is cut into fourths by the hospital pharmacist
  Interventions: Device: misoprostol
- misoprostol and foley bulb group (Active Comparator): Women in the combination group will receive vaginal misoprostol per standard protocol. In addition, a foley bulb will be inserted digitally or by direct visualization with the use of a sterile speculum. The foley will be inserted through the internal os and filled with 60cc of normal saline. The catheter will be taped to the patient's inner thigh under gentle traction. When the foley bulb has fallen out (spontaneous expulsion), further management of labor depends on the labor team. If this does not occur, the catheter will be deflated and removed after 24 hours. Oxytocin will be initiated in those patients who were not in labor after expulsion or removal of the catheter.
  Interventions: Device: misoprostol; Device: Foley bulb

INTERVENTIONS:
Device: misoprostol — 25mcg of misoprostol per vagina every 4hours per the standard hospital protocol. Once the cervix becomes favorable or if the patient is in active labor, or if there is no progress for 24 hours, misoprostol administration will be discontinued. Further management of labor will depend on the labor team. (25mcg tablets are not available commercially; a 100mcg table is cut into fourths by the hospital pharmacist).
  Other Names: cytotec
Device: Foley bulb — a foley bulb will be inserted digitally or by direct visualization with the use of a sterile speculum. The foley will be inserted through the internal os and filled with 60cc of normal saline. The catheter will be taped to the patient's inner thigh under gentle traction. When the foley bulb has fallen out (spontaneous expulsion), further management of labor depends on the labor team. If this does not occur, the catheter will be deflated and removed after 24 hours.
  Other Names: foley bulb (ballon)
  Arms: misoprostol and foley bulb group

SUMMARY:
A randomized, prospective trial will be offered to women admitted to the Roosevelt Hospital labor floor for labor induction. The hypothesis is that the simultaneous use of a foley bulb together with vaginal misoprostol will result in shorter induction to delivery time compared with vaginal misoprostol alone

DETAILED DESCRIPTION:
1. Objectives The hypothesis is that cervical ripening using a foley bulb together with vaginal misoprostol (cytotec) will result in shorter induction to delivery time compared with vaginal misoprostol alone
2. Background The rate of induction of labor in the United States is approximately 20% of all births. Induction of labor can result in prolonged labor and increases the rate of cesarean delivery, both of which are associated with increased maternal and neonatal morbidity. Ripening of an unfavorable cervix has become an integral part of the labor induction process. The best method of cervical ripening remains controversial; no one method has proved to be superior. Women requiring labor induction often present with unfavorable cervices which can lead to a prolonged induction. Cervical ripening is often done to increase the likelihood of successful labor induction.

   Misoprostol (cytotec) is PGE1 analog and widely used for cervical ripening and is the preferred method of induction of labor based on the safety reported literature. Low-dose (25 mcg) intravaginal misoprostol appears to be safe and effective for cervical ripening in term pregnancy for patients without a history of cesarean section. Compared with other cervical ripening methods, misoprostol has an increased rate of vaginal delivery within 24 hours without significant differences in cesarean section rates or fetal outcomes.

   The use of the foley catheter for induction of labor was first described by Krause in 1953. In 1967 Embrey and Mollison reported a 94% successful induction rate after using the foley catheter for cervical ripening. Since then, several studies found transcervical foley catheters as effective as prostaglandins preparations for ripening without an increased risk of uterine rupture.

   There are many proposed methods for induction of labor including mechanical (transcervical foley bulb) and chemical methods (prostaglandins, oxytocin). A number of randomized trials have compared the use of foley bulb, oxytocin and misoprostol in different combinations for induction of labor and their results are contradictory with regards to induction to delivery time, successful vaginal delivery and labor complications.

   There are two studies that evaluated the foley bulb with misoprostol comparing to misoprostol alone. Carbone el al study, found the mean induction to delivery time was 3 hours shorter with the combination of the foley bulb and vaginal misoprostol when compared to vaginal misoprostol alone. In a study by Chung et al, there was no difference in the induction to delivery time.

   Therefore given the contradicting results regarding induction of labor using foley bulb with misoprostol or misoprostol alone, the purpose of our study is to determine if there is a decrease in the induction to delivery time with one method versus the other.
3. Setting of the Human Research Research will take place on the labor and delivery floor of Roosevelt Hospital
4. Study Design a) Recruitment Methods Women admitted to labor and delivery at Roosevelt Hospital will be asked to participate in the study if they are to have an induction of labor at or beyond term (37weeks of gestation). Patients will be screened and those meeting the eligibility criteria will be approached. Informed consent will be obtained.

After a discussion about the study with an eligible interested subject, an investigator will review the consent with them. The investigator will give the potential subject the opportunity to ask any questions and have them answered. Potential participants will be given the opportunity to think about the study. (Only those investigators listed as study personnel and authorized to obtain consent, will obtain informed consent). Once a patient wishes to join the study and informed consent is obtained, the subject can participate. Each subject will receive a signed copy of the consent form. The subject can withdraw from the study at any time without any retribution.

ELIGIBILITY:
Inclusion Criteria

* Term 37 weeks or more, singleton in cephalic presentation
* Age 18 years and older
* Patient admitted for induction of labor

Exclusion Criteria:

* Malpresentation
* Preterm labor less than 37 weeks of gestation
* Patients with fetal anomalies
* Premature rupture of membranes
* If the cervix is closed and unable to place the foley bulb
* Multiple gestation
* Non-reassuring fetal heart tracing
* Contraindication to misoprostol
* Contraindication to vaginal delivery (i.e. placenta previa, vasa previa, active vaginal bleeding, marginal previa, macrosomia, etc). History of prior uterine surgery such as cesarean section or myomectomy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Al-Ibraheemi, MD, Principal Investigator — Mount Sinai St Luke's Roosevelt Hospital
Locations (1):
- Mount Sinai Roosevelt, New York, New York, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Al-Ibraheemi Z, Brustman L, Bimson BE, Porat N, Rosenn B. Misoprostol With Foley Bulb Compared With Misoprostol Alone for Cervical Ripening: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):23-29. doi: 10.1097/AOG.0000000000002403. PMID 29215514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period from September 2015-July 2016, 4767 patients delivered at Mount Sinai West and of these, 1423 deliveries followed induction of labor. A total of 200 patients consented to participate in the study and were randomized, 100 to each group.
Groups:
- Misoprostol Group: 25mcg of misoprostol per vagina every 4hours per the standard hospital protocol. Once the cervix becomes favorable or if the patient is in active labor, or if there is no progress for 24 hours, misoprostol administration will be discontinued. Further management of labor will depend on the labor team. (25mcg tablets are not available commercially; a 100mcg table is cut into fourths by the hospital pharmacist.)
- Misoprostol and Foley Bulb Group: 25mcg of misoprostol per vagina every 4hours per the standard hospital protocol. In addition, a foley bulb will be inserted digitally or by direct visualization with the use of a sterile speculum. The foley will be inserted through the internal os and filled with 60cc of normal saline. The catheter will be taped to the patient's inner thigh under gentle traction. When the foley bulb has fallen out (spontaneous expulsion), further management of labor depends on the labor team. If this does not occur, the catheter will be deflated and removed after 24 hours. Oxytocin will be initiated in those patients who were not in labor after expulsion or removal of the catheter.
Period: Overall Study
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Started | 100 | 100
Completed | 92 | 94
Not Completed | 8 | 6
Not completed — vaginal bleeding | 0 | 1
Not completed — received foley | 8 | 0
Not completed — did not receive foley | 0 | 1
Not completed — labor after randomization | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (5.9) | 31.8 (6.3) | 31.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (6.8) | 31.22 (5.7) | 31.56 (6.3)
Parity [Count of Participants; unit: Participants]
  Nulliparous | 74 | 70 | 144
  Multiparous | 26 | 30 | 56
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 39.4 (1.4) | 39.6 (1.3) | 39.4 (1.4)
Indication for induction [Count of Participants; unit: Participants]
  Oligohydramnios/Polyhydramnios | 21 | 22 | 43
  Post-EDC | 21 | 21 | 42
  Hypertensive disorder | 28 | 20 | 48
  Gestational diabetes/Diabetes | 11 | 11 | 22
  Advanced maternal age | 1 | 4 | 5
  Others | 18 | 22 | 40
Bishop score at misoprostol placement [Mean (Standard Deviation); unit: units on a scale] — 5 item score, each item scored from 0 to 2-3, with total score from 0 to 13. A woman with a low score of 1 would not be expected to go into labor for about 3 weeks. A woman with a higher score of 10 could be expected to go into labor within a few days.
  Also, If the Bishop score is 8 or greater the chances of having a vaginal delivery are good and the cervix is said to be favorable or "ripe" for induction. If the Bishop score is 6 or less the chances of having a vaginal delivery are low and the cervix is said to be unfavorable or "unripe" for induction.
  units on a scale | 2.71 (1.78) | 3.17 (1.94) | 2.9 (1.8)
Mode of delivery [Count of Participants; unit: Participants]
  Spontaneous Vaginal Delivery | 48 | 59 | 107
  Forceps Vaginal Delivery | 2 | 1 | 3
  Vacuum Vaginal Delivery | 12 | 10 | 22
  Cesarean Delivery | 38 | 30 | 68
Indications for cesarean delivery [Count of Participants; unit: Participants] — Population: Only participants who had a Cesarean delivery
  Participants
    Non-reassuring Fetal tracing: number analyzed (Participants) | 38 | 30 | 68
    Non-reassuring Fetal tracing | 20 | 19 | 39
    Arrest of dilation: number analyzed (Participants) | 38 | 30 | 68
    Arrest of dilation | 9 | 6 | 15
    Arrest of descent: number analyzed (Participants) | 38 | 30 | 68
    Arrest of descent | 5 | 4 | 9
    Failed induction of labor: number analyzed (Participants) | 38 | 30 | 68
    Failed induction of labor | 3 | 1 | 4
    Others: number analyzed (Participants) | 38 | 30 | 68
    Others | 1 | 0 | 1
Insurance [Count of Participants; unit: Participants]
  Private | 59 | 53 | 112
  Service | 41 | 47 | 88
Anesthesia [Count of Participants; unit: Participants]
  None | 4 | 6 | 10
  Neuraxial anesthesia | 96 | 91 | 187
  General Anesthesia | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Time Interval From Induction to Delivery: All Participants
Description: During labor from the start of the induction to the delivery
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
hours | 20.97 (10.27) | 16.27 (7.6)

2. Primary Outcome: Time (Hours) From Induction to Delivery: Nulliparous
Time Frame: Day 1
Population: for nulliparous participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 74 | 70
hours | 22.7 (10.58) | 18.15 (7.87)

3. Primary Outcome: Time (Hours) From Induction to Delivery: Multiparous
Time Frame: Day 1
Population: for nulliparous participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 26 | 30
hours | 15.99 (7.4) | 11.89 (4.6)

4. Primary Outcome: Time From Induction to Delivery: VD
Description: Time (hours) from induction to delivery: Vaginal Delivery (VD)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 62 | 70
hours | 18.87 (8) | 15.55 (6.7)

5. Primary Outcome: Time From Induction to Delivery: CD
Description: Time (hours) from induction to delivery: Cesarean Delivery (CD)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 38 | 30
hours | 24.38 (12.49) | 17.95 (9.29)

6. Primary Outcome: Per Treatment Protocol: Time (Hours) From Induction to Delivery
Time Frame: day 1
Population: those participants on treatment protocol
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 92 | 94
hours | 20.5109 (10.09) | 16.6814 (7.47)

7. Secondary Outcome: The Time From Induction Until to Active Phase Labor
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
hours | 17.43 (8.6) | 12.81 (5.83)

8. Secondary Outcome: The Time From Active Phase to Delivery
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
hours | 3.11 (2.75) | 3.76 (3)

9. Secondary Outcome: Incidence of Chorioamnionitis
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
Participants | 8 | 4

10. Secondary Outcome: Incidence of Uterine Tachysystole
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
Participants | 12 | 6

11. Secondary Outcome: Incidence of Patient Discomfort
Time Frame: Day 1
Population: data not collected
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Estimated Blood Loss
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
Number analyzed (Participants) | 100 | 100
ml | 493.3 (274) | 490.5 (304.1)

ADVERSE EVENTS:
Arm/Group | Misoprostol Group | Misoprostol and Foley Bulb Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes